CLINICAL TRIAL: NCT07401979
Title: The Influence of Explainability and Integrability of AI-CDSS on Usage Behavior Among Primary Care Physicians
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yushu Liu, Principal Investigator, Huazhong University of Science and Technology
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: CXL202601141106
Record Dates: First submitted 2026-01-19; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Respiratory Tract Infections (RTI)
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (32):
- AI-CDSS Basic Configuration (No Intervention): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (disabled), Confidence Display (disabled), Feature Importance (disabled), Stepwise Medication (disabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
- AI-CDSS Configuration 2 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (disabled), Confidence Display (disabled), Feature Importance (disabled), Stepwise Medication (enabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with Stepwise Medication and Auto-extraction
- AI-CDSS Configuration 3 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (disabled), Confidence Display (disabled), Feature Importance (enabled), Stepwise Medication (disabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with Feature Importance and Auto-extraction
- AI-CDSS Configuration 4 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (disabled), Confidence Display (disabled), Feature Importance (enabled), Stepwise Medication (enabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with Feature Importance and Stepwise Medication
- AI-CDSS Configuration 5 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (disabled), Confidence Display (enabled), Feature Importance (disabled), Stepwise Medication (disabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with Confidence Display and Auto-extraction
- AI-CDSS Configuration 6 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (disabled), Confidence Display (enabled), Feature Importance (disabled), Stepwise Medication (enabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with Confidence Display and Stepwise Medication
- AI-CDSS Configuration 7 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (disabled), Confidence Display (enabled), Feature Importance (enabled), Stepwise Medication (disabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with Confidence Display and Feature Importance
- AI-CDSS Configuration 8 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (disabled), Confidence Display (enabled), Feature Importance (enabled), Stepwise Medication (enabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with 4 Features (Config 8)
- AI-CDSS Configuration 9 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (enabled), Confidence Display (disabled), Feature Importance (disabled), Stepwise Medication (disabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with Chain-of-Thought Reasoning and Auto-extraction
- AI-CDSS Configuration 10 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (enabled), Confidence Display (disabled), Feature Importance (disabled), Stepwise Medication (enabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with Chain-of-Thought Reasoning and Stepwise Medication
- AI-CDSS Configuration 11 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (enabled), Confidence Display (disabled), Feature Importance (enabled), Stepwise Medication (disabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with Chain-of-Thought Reasoning and Feature Importance
- AI-CDSS Configuration 12 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (enabled), Confidence Display (disabled), Feature Importance (enabled), Stepwise Medication (enabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with 4 Features (Config 12)
- AI-CDSS Configuration 13 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (enabled), Confidence Display (enabled), Feature Importance (disabled), Stepwise Medication (disabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with Chain-of-Thought Reasoning and Confidence Display
- AI-CDSS Configuration 14 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (enabled), Confidence Display (enabled), Feature Importance (disabled), Stepwise Medication (enabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with 4 Features (Config 14)
- AI-CDSS Configuration 15 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (enabled), Confidence Display (enabled), Feature Importance (enabled), Stepwise Medication (disabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with 4 Features (Config 15)
- AI-CDSS Configuration 16 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (disabled), Chain-of-Thought Reasoning (enabled), Confidence Display (enabled), Feature Importance (enabled), Stepwise Medication (enabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with 4 Features (Config 16)
- AI-CDSS Configuration 17 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (disabled), Confidence Display (disabled), Feature Importance (disabled), Stepwise Medication (disabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with Sidebar Display and Auto-extraction
- AI-CDSS Configuration 18 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (disabled), Confidence Display (disabled), Feature Importance (disabled), Stepwise Medication (enabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with Sidebar Display and Stepwise Medication
- AI-CDSS Configuration 19 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (disabled), Confidence Display (disabled), Feature Importance (enabled), Stepwise Medication (disabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with Sidebar Display and Feature Importance
- AI-CDSS Configuration 20 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (disabled), Confidence Display (disabled), Feature Importance (enabled), Stepwise Medication (enabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with 4 Features (Config 20)
- AI-CDSS Configuration 21 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (disabled), Confidence Display (enabled), Feature Importance (disabled), Stepwise Medication (disabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with Sidebar Display and Confidence Display
- AI-CDSS Configuration 22 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (disabled), Confidence Display (enabled), Feature Importance (disabled), Stepwise Medication (enabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with 4 Features (Config 22)
- AI-CDSS Configuration 23 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (disabled), Confidence Display (enabled), Feature Importance (enabled), Stepwise Medication (disabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with 4 Features (Config 23)
- AI-CDSS Configuration 24 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (disabled), Confidence Display (enabled), Feature Importance (enabled), Stepwise Medication (enabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with 4 Features (Config 24)
- AI-CDSS Configuration 25 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (enabled), Confidence Display (disabled), Feature Importance (disabled), Stepwise Medication (disabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with Sidebar Display and Chain-of-Thought Reasoning
- AI-CDSS Configuration 26 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (enabled), Confidence Display (disabled), Feature Importance (disabled), Stepwise Medication (enabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with 4 Features (Config 26)
- AI-CDSS Configuration 27 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (enabled), Confidence Display (disabled), Feature Importance (enabled), Stepwise Medication (disabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with 4 Features (Config 27)
- AI-CDSS Configuration 28 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (enabled), Confidence Display (disabled), Feature Importance (enabled), Stepwise Medication (enabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with 4 Features (Config 28)
- AI-CDSS Configuration 29 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (enabled), Confidence Display (enabled), Feature Importance (disabled), Stepwise Medication (disabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with 4 Features (Config 29)
- AI-CDSS Configuration 30 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (enabled), Confidence Display (enabled), Feature Importance (disabled), Stepwise Medication (enabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with 4 Features (Config 30)
- AI-CDSS Configuration 31 (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (enabled), Confidence Display (enabled), Feature Importance (enabled), Stepwise Medication (disabled), Auto-extraction (disabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: AI-CDSS with 4 Features (Config 31)
- AI-CDSS Full Configuration (Experimental): Participants interact with an AI Clinical Decision Support System with the following feature settings: Sidebar Display (enabled), Chain-of-Thought Reasoning (enabled), Confidence Display (enabled), Feature Importance (enabled), Stepwise Medication (enabled), Auto-extraction (enabled). Participants complete 3 clinical case evaluations for respiratory tract infections using this AI configuration.
  Interventions: Behavioral: Full-Featured AI-CDSS

INTERVENTIONS:
Behavioral: AI-CDSS with Stepwise Medication and Auto-extraction — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Stepwise Medication; Auto-extraction. Inactive features: Sidebar Display; Chain-of-Thought Reasoning; Confidence Display; Feature Importance. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 2
Behavioral: AI-CDSS with Feature Importance and Auto-extraction — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Feature Importance; Auto-extraction. Inactive features: Sidebar Display; Chain-of-Thought Reasoning; Confidence Display; Stepwise Medication. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 3
Behavioral: AI-CDSS with Feature Importance and Stepwise Medication — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Feature Importance; Stepwise Medication. Inactive features: Sidebar Display; Chain-of-Thought Reasoning; Confidence Display; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 4
Behavioral: AI-CDSS with Confidence Display and Auto-extraction — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Confidence Display; Auto-extraction. Inactive features: Sidebar Display; Chain-of-Thought Reasoning; Feature Importance; Stepwise Medication. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 5
Behavioral: AI-CDSS with Confidence Display and Stepwise Medication — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Confidence Display; Stepwise Medication. Inactive features: Sidebar Display; Chain-of-Thought Reasoning; Feature Importance; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 6
Behavioral: AI-CDSS with Confidence Display and Feature Importance — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Confidence Display; Feature Importance. Inactive features: Sidebar Display; Chain-of-Thought Reasoning; Stepwise Medication; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 7
Behavioral: AI-CDSS with 4 Features (Config 8) — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Confidence Display; Feature Importance; Stepwise Medication; Auto-extraction. Inactive features: Sidebar Display; Chain-of-Thought Reasoning. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 8
Behavioral: AI-CDSS with Chain-of-Thought Reasoning and Auto-extraction — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Chain-of-Thought Reasoning; Auto-extraction. Inactive features: Sidebar Display; Confidence Display; Feature Importance; Stepwise Medication. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 9
Behavioral: AI-CDSS with Chain-of-Thought Reasoning and Stepwise Medication — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Chain-of-Thought Reasoning; Stepwise Medication. Inactive features: Sidebar Display; Confidence Display; Feature Importance; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 10
Behavioral: AI-CDSS with Chain-of-Thought Reasoning and Feature Importance — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Chain-of-Thought Reasoning; Feature Importance. Inactive features: Sidebar Display; Confidence Display; Stepwise Medication; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 11
Behavioral: AI-CDSS with 4 Features (Config 12) — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Chain-of-Thought Reasoning; Feature Importance; Stepwise Medication; Auto-extraction. Inactive features: Sidebar Display; Confidence Display. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 12
Behavioral: AI-CDSS with Chain-of-Thought Reasoning and Confidence Display — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Chain-of-Thought Reasoning; Confidence Display. Inactive features: Sidebar Display; Feature Importance; Stepwise Medication; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 13
Behavioral: AI-CDSS with 4 Features (Config 14) — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Chain-of-Thought Reasoning; Confidence Display; Stepwise Medication; Auto-extraction. Inactive features: Sidebar Display; Feature Importance. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 14
Behavioral: AI-CDSS with 4 Features (Config 15) — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Chain-of-Thought Reasoning; Confidence Display; Feature Importance; Auto-extraction. Inactive features: Sidebar Display; Stepwise Medication. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 15
Behavioral: AI-CDSS with 4 Features (Config 16) — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Chain-of-Thought Reasoning; Confidence Display; Feature Importance; Stepwise Medication. Inactive features: Sidebar Display; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 16
Behavioral: AI-CDSS with Sidebar Display and Auto-extraction — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Auto-extraction. Inactive features: Chain-of-Thought Reasoning; Confidence Display; Feature Importance; Stepwise Medication. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 17
Behavioral: AI-CDSS with Sidebar Display and Stepwise Medication — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Stepwise Medication. Inactive features: Chain-of-Thought Reasoning; Confidence Display; Feature Importance; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 18
Behavioral: AI-CDSS with Sidebar Display and Feature Importance — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Feature Importance. Inactive features: Chain-of-Thought Reasoning; Confidence Display; Stepwise Medication; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 19
Behavioral: AI-CDSS with 4 Features (Config 20) — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Feature Importance; Stepwise Medication; Auto-extraction. Inactive features: Chain-of-Thought Reasoning; Confidence Display. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 20
Behavioral: AI-CDSS with Sidebar Display and Confidence Display — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Confidence Display. Inactive features: Chain-of-Thought Reasoning; Feature Importance; Stepwise Medication; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 21
Behavioral: AI-CDSS with 4 Features (Config 22) — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Confidence Display; Stepwise Medication; Auto-extraction. Inactive features: Chain-of-Thought Reasoning; Feature Importance. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 22
Behavioral: AI-CDSS with 4 Features (Config 23) — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Confidence Display; Feature Importance; Auto-extraction. Inactive features: Chain-of-Thought Reasoning; Stepwise Medication. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 23
Behavioral: AI-CDSS with 4 Features (Config 24) — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Confidence Display; Feature Importance; Stepwise Medication. Inactive features: Chain-of-Thought Reasoning; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 24
Behavioral: AI-CDSS with Sidebar Display and Chain-of-Thought Reasoning — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Chain-of-Thought Reasoning. Inactive features: Confidence Display; Feature Importance; Stepwise Medication; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 25
Behavioral: AI-CDSS with 4 Features (Config 26) — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Chain-of-Thought Reasoning; Stepwise Medication; Auto-extraction. Inactive features: Confidence Display; Feature Importance. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 26
Behavioral: AI-CDSS with 4 Features (Config 27) — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Chain-of-Thought Reasoning; Feature Importance; Auto-extraction. Inactive features: Confidence Display; Stepwise Medication. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 27
Behavioral: AI-CDSS with 4 Features (Config 28) — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Chain-of-Thought Reasoning; Feature Importance; Stepwise Medication. Inactive features: Confidence Display; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 28
Behavioral: AI-CDSS with 4 Features (Config 29) — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Chain-of-Thought Reasoning; Confidence Display; Auto-extraction. Inactive features: Feature Importance; Stepwise Medication. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 29
Behavioral: AI-CDSS with 4 Features (Config 30) — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Chain-of-Thought Reasoning; Confidence Display; Stepwise Medication. Inactive features: Feature Importance; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 30
Behavioral: AI-CDSS with 4 Features (Config 31) — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Chain-of-Thought Reasoning; Confidence Display; Feature Importance. Inactive features: Stepwise Medication; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Configuration 31
Behavioral: Full-Featured AI-CDSS — An artificial intelligence-based Clinical Decision Support System for respiratory tract infections. Active features: Sidebar Display; Chain-of-Thought Reasoning; Confidence Display; Feature Importance; Stepwise Medication; Auto-extraction. The system provides diagnosis suggestions and antibiotic recommendations for primary care physicians.
  Arms: AI-CDSS Full Configuration

SUMMARY:
The goal of this observational experimental study is to determine how system-level features of artificial intelligence clinical decision support systems (AI-CDSS)-specifically explainability and integrability-affect usage behavior among primary care physicians in China. The study focuses on licensed primary care physicians, regardless of gender, age, years of clinical experience, or prior AI exposure.

The main questions it aims to answer are:

* Do specific AI features (e.g., feature attribution, chain-of-thought explanation, seamless workflow integration, automated data input) independently influence physicians' adoption intention, diagnostic accuracy, and their perceptions of the system's usefulness and ease of use?
* Do pairwise combinations of these AI features produce significant interaction effects-either synergistic or antagonistic-on these outcomes? Researchers will compare 32 distinct AI interface configurations generated from a 2⁶-¹ fractional factorial design (Resolution VI), each representing a unique combination of six binary AI features: (A) gradient-based feature importance (0 = absent, 1 = present), (B) chain-of-thought reasoning (0/1), (C) workflow integration (0 = multiple pop-up alerts, 1 = unified sidebar display), (D) automated data extraction (0 = manual entry, 1 = auto-populated from case text), (E) recommendation scope adapted to primary care settings (0 = restricted to essential options, 1 = full range of recommendations), and (F) model confidence display (0 = absent, 1 = present). This design enables unbiased estimation of all six main effects and all 15 two-way interactions.

Participants will:

Complete three standardized clinical case scenarios involving common respiratory infections via a web-based simulation platform; First provide an initial diagnosis and treatment plan without any AI input; Then review an AI-generated recommendation embedded with a randomly assigned combination of the six AI features; Revise their final diagnosis and prescription based on the AI suggestion; Rate their adoption intention, perceived usefulness, and perceived ease of use using validated 7-point Likert-scale items after each case.

ELIGIBILITY:
Inclusion Criteria:

1. Be currently employed full-time in clinical practice at a primary care facility, including community health centers, community health stations, township hospitals, or village clinics;
2. Hold a clinical medical license with a specialty in general practice or internal medicine, and have experience in diagnosing and managing respiratory tract infections;
3. Have at least one year of clinical work experience;
4. Be proficient in basic computer use (e.g., web browsing and online questionnaire completion), have reliable internet access, and be capable of independently completing the online experimental tasks;
5. Provide voluntary informed consent to participate in the study.

Exclusion Criteria:

1. Non-clinical staff (e.g., administrative personnel, pharmacists, laboratory technicians, or public health workers who do not directly provide outpatient clinical care);
2. Individuals unable to independently complete the online experimental procedure or who demonstrate significant difficulty understanding the task instructions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Correction Event Rate | Immediately after intervention
  Proportion of cases where the physician's initial decision was incorrect, but was corrected to the right decision after viewing AI recommendations. Calculated as: (Number of cases where initial decision was wrong AND final decision was correct) / (Total number of cases where initial decision was wrong). This measures the positive corrective influence of AI-CDSS on physician decision-making. Continuous variable ranging from 0 to 1.
Misleading Event Rate | Immediately after intervention
  Proportion of cases where the physician's initial decision was correct, but was changed to an incorrect decision after viewing AI recommendations. Calculated as: (Number of cases where initial decision was correct AND final decision was wrong) / (Total number of cases where initial decision was correct). This measures the potential negative influence of AI-CDSS on physician decision-making. Continuous variable ranging from 0 to 1.
Diagnostic Accuracy (Top-1) | Immediately after intervention
  Proportion of cases where the physician's final primary diagnosis (first-ranked diagnosis) matches the correct diagnosis (gold standard). Measured separately for initial diagnosis (before AI) and final diagnosis (after AI) to assess AI impact on diagnostic accuracy. Continuous variable ranging from 0 to 1.
Diagnostic Accuracy (Top-3) | Immediately after intervention
  Proportion of cases where the correct diagnosis (gold standard) appears within the physician's top 3 differential diagnoses. Measured separately for initial diagnosis (before AI) and final diagnosis (after AI). This captures whether the correct diagnosis was considered even if not ranked first. Continuous variable ranging from 0 to 1.
Appropriateness of Antibiotic Use Decision | Immediately after intervention
  Proportion of cases where the physician's final decision on whether to prescribe antibiotics (yes/no) aligns with evidence-based guidelines (gold standard). This measures the appropriateness of the binary decision to use or withhold antibiotics, regardless of the specific antibiotic chosen. Measured separately for initial decision (before AI) and final decision (after AI). Continuous variable ranging from 0 to 1.
Appropriateness of Antibiotic Selection | Immediately after intervention
  Among cases where antibiotics were prescribed, proportion of cases where the physician's final antibiotic selection (specific drug choice) aligns with evidence-based guidelines (gold standard). This measures the appropriateness of the specific antibiotic chosen, conditional on the decision to prescribe. Measured separately for initial selection (before AI) and final selection (after AI). Continuous variable ranging from 0 to 1.

SECONDARY OUTCOMES:
Decision Certainty | Immediately after intervention
  Physician's self-reported confidence level in their final clinical decision after viewing AI recommendations. Measured using a 5-point Likert scale: 1 = Very Uncertain, 2 = Uncertain, 3 = Neutral, 4 = Certain, 5 = Very Certain. This reflects the cognitive impact of AI-CDSS on decision confidence.
Intention to Adopt AI-CDSS | Immediately after intervention
  Measured using a 3-item scale adapted from the Technology Acceptance Model (TAM). Items assess: (1) willingness to apply AI-CDSS in daily clinical practice when available, (2) intention to use AI-CDSS based on actual patient care needs, and (3) willingness to frequently use AI-CDSS when conditions permit. Each item is rated on a 5-point Likert scale (1=Strongly Disagree to 5=Strongly Agree). Total score ranges from 3 to 15.
Perceived Usefulness of AI-CDSS | Immediately after intervention
  Measured using a 6-item Perceived Usefulness scale adapted from TAM (Davis, 1989). Items assess perceived improvements in: (1) task completion speed, (2) job performance, (3) productivity, (4) work effectiveness, (5) ease of work, and (6) overall usefulness. Each item is rated on a 7-point Likert scale (1=Strongly Disagree to 7=Strongly Agree). Total score ranges from 6 to 42.
Perceived Ease of Use of AI-CDSS | Immediately after intervention
  Measured using a 6-item Perceived Ease of Use scale adapted from TAM (Davis, 1989). Items assess: (1) ease of learning, (2) ease of getting desired functions, (3) clarity of interaction, (4) flexibility of interaction, (5) ease of becoming proficient, and (6) overall ease of use. Each item is rated on a 7-point Likert scale (1=Strongly Disagree to 7=Strongly Agree). Total score ranges from 6 to 42.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Medical College of Huazhong University of Science & Technology School of Medicine and Health Management, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No